CLINICAL TRIAL: NCT06110286
Title: Comparison of Corneal High Order Aberrations After Stream Light Trans-PRK and Mechanical Photorefractive Keratectomy
Brief Title: Corneal High Order Aberrations After Stream Light and Mechanical Photorefractive Keratectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate professor, Assiut University
Other Study IDs: 1799
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Compare Corneal High Order Aberrations Before and After Stream Light Trans-PRK and Mechanical Photorefractive Keratectomy
MeSH Terms: interventions — Photorefractive Keratectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Mechanical photorefractive keratectomy: Laser photorefractive keratecyomy by Ex500 excimer laser after mannual removal of corneal epithelium
  Interventions: Other: Photorefractive keratectomy
- Stream light trans-PRK: Laser photorefractive keratectomy by Ex500 excimer laser after removal of corneal epithelium by stream-light laser technique
  Interventions: Other: Photorefractive keratectomy

INTERVENTIONS:
Other: Photorefractive keratectomy — Laser keratectomy by EX500 excimer laser after removal of corneal epithelium either mannually or by laser ablation

SUMMARY:
Compare corneal high order aberrations before and after stream light trans-PRK and mechanical photorefractive keratectomy including third order aberrations; Trefoil and coma aberrations and forth order aberrations; spherical aberrations

DETAILED DESCRIPTION:
Laser technology has played an important role in promoting the development of ophthalmology, especially corneal refractive surgery.1 Trans-epithelial photorefractive keratectomy (Trans-PRK) has become a highly researched topic in recent years.2 Different epithelial debridement methods with PRK showed favorable results for the surgical treatment of low to moderate myopia3. In mechanical PRK (m-PRK), epithelial debridement is achieved using a blunt spatula, whereas in stream light trans-PRK (t-PRK), there after an excimer laser is used to ablate corneal stroma3. The Stream Light t-PRK is a safe and effective treatment option for the correction of low to moderate myopia.4 Many studies have shown that the corneal asphericity developed significantly after refractive surgeries and introduce higher-order aberrations (HOAs).2 The present study focused on three of the most clinically important HOAs; spherical, coma, and trefoil aberrations, both preoperative and postoperative were recorded from topography over the 6-mm-diameter central corneal zone using Pentacam.

ELIGIBILITY:
Inclusion Criteria:

* • Stable refraction for 1 year (refraction does not exceed 1D more than the last prescribed glasses).

  * Discontinuation of soft contact lens wears at least 1 week before examination.
  * Topography criteria:
* Corneal thickness equal or more than 470 um
* Symmetrical bow-tie
* Back elevation not more than +12
* Normal Belin\Ambrosio Enhanced ectasia display
* Spherical equivalent not more than -6D.

Exclusion Criteria:

* • Previous ocular surgery

  * Concurrent ocular pathology; corneal scar, corneal dystrophy
  * Systemic disease; Uncontrolled diabetes, collagen disease
  * Post-operative complications; sub-epithelial haze.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Myopic patients with spherical equivalent not more than -6D who will present to refractive surgery Centre in Assiut and seeking for refractive surgery to get rid of their glasses and fulfilling the inclusion and exclusion criteria
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Corneal high order aberrations measured before and after the intervention by corneal topography machine | 1 monthe after surgery
  * Third order aberrations; Trefoil and coma aberrations
  * Forth order aberrations; spherical aberrations Trefoil, spherical and coma aberrations

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university faculty of medicine, Asyut, Assiut University, Egypt